CLINICAL TRIAL: NCT07201272
Title: Ultrasound-Guided Transversalis Fascia Plane Block Versus Intrathecal Morphine for Postoperative Analgesia in Patients Undergoing Total Abdominal Hysterectomy: A Randomized Clinical Trial
Brief Title: Transversalis Fascia Plane Block Versus Intrathecal Morphine for Postoperative Analgesia in Total Abdominal Hysterectomy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Mohammed Said ElSharkawy, Lecturer of Anesthesiology, Surgical Intensive Care and Pain Medicine, Faculty of Medicine, Tanta University, Tanta, Egypt., Tanta University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 36264PR1337/8/25
Record Dates: First submitted 2025-09-23; First posted 2025-10-01 (Actual); Last update posted 2025-10-02 (Actual); Status verified 2025-10

CONDITIONS: Transversalis Fascia Plane Block; Intrathecal Morphine; Postoperative Analgesia; Total Abdominal Hysterectomy
MeSH Terms: interventions — Morphine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- TFP group (Experimental): Patients will receive spinal anesthesia (using 3.5 mL of hyperbaric bupivacaine 0.5%) with bilateral transversalis fascia plane (TFP) block (using 20 mL of bupivacaine 0.25%) at the end of surgery.
  Interventions: Other: Transversalis fascia plane block
- IM group (Experimental): Patients will receive spinal anesthesia (using 3 mL of hyperbaric bupivacaine 0.5%) + (75 µg morphine diluted in 0.5ml saline) with sham block at the end of surgery.
  Interventions: Drug: Morphine

INTERVENTIONS:
Other: Transversalis fascia plane block — Patients will receive spinal anesthesia (using 3.5 mL of hyperbaric bupivacaine 0.5%) with bilateral transversalis fascia plane (TFP) block (using 20 mL of bupivacaine 0.25%) at the end of surgery.
  Arms: TFP group
Drug: Morphine — Patients will receive spinal anesthesia (using 3 mL of hyperbaric bupivacaine 0.5%) + (75 µg morphine diluted in 0.5ml saline) with sham block at the end of surgery.
  Arms: IM group

SUMMARY:
This study aims to compare the ultrasound-guided transversalis fascia plane (TFP) block and intrathecal morphine for postoperative analgesia in patients undergoing total abdominal hysterectomy (TAH).

DETAILED DESCRIPTION:
Total abdominal hysterectomy (TAH) is a commonly performed major surgical procedure that results in substantial postoperative pain and discomfort. Postoperative pain, if not treated promptly, can impair the patient's ability to ambulate which may lead to adverse effects such as thromboembolism, myocardial ischemia, and arrhythmia.

Intrathecal opioids are synergistic with local anesthetics and intensify the sensory block without increasing the sympathetic block. Morphine, which is relatively less hydrophobic than other opioids, has a longer residence time in the cerebrospinal fluid and therefore may reach rostral sites over a longer period than other opioids.

Ultrasound-guided interfascial plane blocks are often used in multimodal analgesia regimens. Local anaesthetic injection into the transversalis fascia plane (TFP) anesthetizes the proximal branches of T12 and L1 which targeted in the plane between the transversus abdominis muscle and the transversalis fascia.

ELIGIBILITY:
Inclusion Criteria:

* Age from 18 to 65 years.
* American Society of Anesthesiology (ASA) physical status I-II.
* Women undergoing total abdominal hysterectomy (TAH) under spinal anesthesia.

Exclusion Criteria:

* History of allergies to local anesthetics.
* Local infection at the site of injection.
* Bleeding disorders.
* History of chronic use of analgesic.
* Physical or mental conditions.
* Hepatic, renal or cardiac disease.
* Contraindication to spinal anesthesia.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Women Undergoing Total Abdominal Hysterectomy
Enrollment: 60 (Estimated)
Dates: Start 2025-10-01 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
Time to the 1st rescue analgesia | 24 hours postoperatively
  Time to the first request for the rescue analgesia (time from the end of surgery to first dose of morphine administrated).

SECONDARY OUTCOMES:
Total morphine consumption | 24 hours postoperatively
  Rescue analgesia of morphine will be given as 3 mg bolus if the numeric rating scale (NRS)> 3 to be repeated after 30 min if pain persists until the NRS < 4.
Degree of pain | 24 hours postoperatively
  Each patient will be instructed about postoperative pain assessment with the numeric rating scale (NRS). NRS (0 represents "no pain" while 10 represents "the worst pain imaginable"). NRS will be assessed at post-anesthesia care unit (PACU), 2, 4, 6, 8, 12, 18, and 24 h postoperatively.
Incidence of adverse events | 24 hours postoperatively
  Incidence of adverse events such as bradycardia, hypotension, pruritis, nausea, vomiting, respiratory depression, or any other complication will be recorded.

CONTACTS AND LOCATIONS:
Locations (1):
- Tanta University, Tanta, Egypt

IPD SHARING:
Plan to Share IPD: Yes
The data will be available upon a reasonable request from the corresponding author after the end of study for one year.
Supporting Information: Study Protocol
Time Frame: After the end of study for one year.
Access Criteria: The data will be available upon a reasonable request from the corresponding author.